CLINICAL TRIAL: NCT05892341
Title: A Clinical Study to Compare the Performance of AQUACEL® Ag+ Extra™ and Cutimed® Sorbact® Dressing in the Management of Patients With Venous Leg Ulcers Over a 12-week Period
Brief Title: AQUACEL® Ag+ Extra™ and Cutimed™ Sorbact® Dressing in the Management of Venous Leg Ulcers Over a 12-week Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WC-22-435
Record Dates: First submitted 2023-05-10; First posted 2023-06-07 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Venous Leg Ulcer; Diabetic Foot
MeSH Terms: conditions — Varicose Ulcer; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AQUACEL® Ag+ Extra™ (Active Comparator): AQUACEL® Ag+ Extra™ is approved, needle-bonded nonwoven fabric layered and stitch-bonded wound dressing
  Interventions: Device: AQUACEL® Ag+ Extra™
- Cutimed® Sorbact® (Active Comparator): Cutimed® Sorbact® is approved, bacterial and fungi binding wound dressing
  Interventions: Device: Cutimed® Sorbact®

INTERVENTIONS:
Device: AQUACEL® Ag+ Extra™ — Wound treatment with AQUACEL® Ag+ Extra™ dressing
  Arms: AQUACEL® Ag+ Extra™
Device: Cutimed® Sorbact® — Wound treatment with Cutimed® Sorbact® dressing
  Arms: Cutimed® Sorbact®

SUMMARY:
Study is to provide evidence comparing AQUACEL® Ag+ Extra™ versus Cutimed® Sorbact® in the progression of wounds towards healing

DETAILED DESCRIPTION:
Post market, multi-centre, randomised, open label, multi-national, prospective study to provide evidence comparing AQUACEL® Ag+ Extra™ versus Cutimed® Sorbact® in the progression of wounds towards healing

ELIGIBILITY:
Inclusion Criteria:

* Venous insufficiency as defined by CEAP Classification of C6
* One wound amendable to treatment with either AQUACEL® Ag+ Extra™ or Cutimed® Sorbact®
* Wounds that have been present for at least 2 months
* Reliable and available for follow-up
* 18 years or older
* Able and willing to provide informed consent
* Able to tolerate compression therapy for Venus Leg Ulcer
* Must be able to be compliant with compression therapy

Exclusion Criteria:

* Known sensitivities or allergies to components of the AQUACEL® Ag+ Extra™ or Cutimed® Sorbact®
* Continued use of petroleum gel/ creams/ oil-based products
* Active treatment for cancer or completed within the last 3 months
* Documented severe malnutrition
* Malignant wounds
* Systemic infection actively treated with antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Saavedra, MD, Principal Investigator — Convatec Colombia Clinic
Locations (18):
- Colombia (6):
  - Convatec Colombia Clinic, Barranquilla
  - Convatec Colombia Clinic, Bogotá
  - Convatec Colombia Clinic, Bucaramanga
  - Convatec Colombia Clinic, Cali
  - Convatec Colombia Clinic, Cartagena
  - Convatec Colombia Clinic, Medellín
- Germany (11):
  - Germany, Augsburg
  - Germany, Berlin
  - Germany, Bochum
  - Germany, Düsseldorf
  - Germany, Holzkirchen
  - Germany, Ingolstadt
  - Germany Clinic II, München
  - Germany Clinic I, München
  - Germany, Nuremberg
  - Germany, Ratzeburg
  - Germany, Rosenheim
- VCTC UK, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Wounds
Period: Overall Study
Arm/Group | AQUACEL® Ag+ Extra™ | Cutimed® Sorbact®
Started | 101; 109 Wounds | 102; 110 Wounds
Completed | 88; 96 Wounds | 79; 85 Wounds
Not Completed | 13; 13 Wounds | 23; 25 Wounds

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AQUACEL® Ag+ Extra™ | Cutimed® Sorbact® | Total
Number analyzed (Participants) | 101 | 102 | 203
Age, Customized [Count of Participants; unit: Participants] — Age years, Categorical
  Participants
    < 65 | 38 | 42 | 80
    65-79 | 44 | 41 | 85
    80+ | 19 | 19 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 56 | 127
  Male | 30 | 46 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Colombia | 59 | 59 | 118
  United Kingdom | 20 | 22 | 42
  Germany | 22 | 21 | 43
BMI [Mean (Standard Deviation); unit: kg/m2] | 31.84 (8.26) | 30.06 (6.12) | 30.95 (7.19)

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of AQUACEL® Ag+ Extra™ and Cutimed® Sorbact® on Wound Management
Description: Complete wound closure as defined by 100% epithelialisation of the wound surface (Gould 2019)
Time Frame: Up to 12 weeks
Population: Proportion of study wounds with complete wound healing by Week 12
Measure: Count of Units; unit: Number of Wounds
Units Other Than Participants: Number of Wounds
Arm/Group | AQUACEL® Ag+ Extra™ | Cutimed® Sorbact®
Number analyzed (Participants) | 101 | 102
Number analyzed (Number of Wounds) | 107 | 108
Number of Wounds | 80 | 60

2. Secondary Outcome: Wound Healing Assessment
Description: Percent change in study wound area
Time Frame: Up to 4 weeks
Population: Percent change in wound size at Week 4
Measure: Mean (Standard Deviation); unit: Percent change in wound size
Units Other Than Participants: Number of Wounds
Arm/Group | AQUACEL® Ag+ Extra™ | Cutimed® Sorbact®
Number analyzed (Participants) | 101 | 102
Number analyzed (Number of Wounds) | 105 | 108
Percent change in wound size | -62.66 (43.54) | -48.31 (49.97)

3. Secondary Outcome: Wound Progress Assessment
Description: Satisfactory clinical progress defined as 40% reduction in study wound area
Time Frame: Up to 4 weeks
Population: Proportion of study wounds with satisfactory clinical progress defined as 40% reduction in study wound area at 4 weeks
Measure: Number (95% Confidence Interval); unit: Number of Wounds
Units Other Than Participants: Number of Wounds
Arm/Group | AQUACEL® Ag+ Extra™ | Cutimed® Sorbact®
Number analyzed (Participants) | 101 | 102
Number analyzed (Number of Wounds) | 105 | 108
Number of Wounds | 81 [69.11 to 85.17] | 70 [55.81 to 73.82]

4. Secondary Outcome: Wound Change Assessment
Description: Percent change in target wound area
Time Frame: Up to 12 weeks
Population: Percent change in wound size at Week 12
Measure: Mean (Standard Deviation); unit: Percent change in wound size
Units Other Than Participants: Number of Wounds
Arm/Group | AQUACEL® Ag+ Extra™ | Cutimed® Sorbact®
Number analyzed (Participants) | 101 | 102
Number analyzed (Number of Wounds) | 105 | 108
Percent change in wound size | -90.33 (27.09) | -67.22 (55.13)

5. Secondary Outcome: Safety Assesment
Description: Summary of the incidence of adverse events (AEs), device-related adverse events (ADEs) and serious device-related adverse events (SADEs)
Time Frame: Up to 12 weeks
Population: Proportion of subjects with AEs, SAEs, ADEs and Unanticipated Adverse Device Effects
Measure: Number; unit: participants
Arm/Group | AQUACEL® Ag+ Extra™ | Cutimed® Sorbact®
Number analyzed (Participants) | 101 | 102
participants
  Any AE, subjects | 11 | 27
  Any SAE, subjects | 3 | 6
  Adverse Device Effects | 1 | 4
  Serious Adverse Device Effect | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs), Serious Adverse events (SAEs), Adverse Device Effects (ADEs), Serious Adverse Device Effects (SADEs), Unanticipated Serious Adverse Device Effects (UADEs) and Device deficiencies were recorded throughout the study duration up to 84 days (±2 days).
Description: The definitions of each type of these events, instructions for causality assessment (i.e., determination of relationship of the event to the study device or study procedure), categories of severity (mild, moderate, or severe) of events, and procedure for monitoring and recording of events were provided in the study Protocol.
Arm/Group | AQUACEL® Ag+ Extra™ | Cutimed® Sorbact®
All-Cause Mortality (participants affected / at risk) | 0/101 | 1/102
Serious Adverse Events (participants affected / at risk) | 3/101 | 6/102
Other Adverse Events (participants affected / at risk) | 8/101 | 21/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AQUACEL® Ag+ Extra™ (N=101) | Cutimed® Sorbact® (N=102)
Ischaemic heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Allergic reaction to drug (Immune system disorders) | 0 (0) | 1 (1)
Cellulitis on left lower leg (Infections and infestations) | 0 (0) | 1 (1)
Chest infection (Infections and infestations) | 1 (1) | 0 (0)
UTI (Infections and infestations) | 1 (1) | 1 (1)
Unspecified local infection of skin and subcutaneous tissue (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AQUACEL® Ag+ Extra™ (N=101) | Cutimed® Sorbact® (N=102)
Wound infection (Infections and infestations) | 3 (3) | 4 (4)
UTI (Infections and infestations) | 1 (1) | 0 (0)
Ulcer bleeding (General disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overgranulation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Unilateral leg swelling (General disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Thrush (Infections and infestations) | 0 (0) | 1 (1)
Thumb osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Leg ulcer (not study ulcer) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Wound pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) — Increase in pain associated with right leg ulcer
Open wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Open wound great toe right foot
Itching all over (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ulcer (General disorders) | 1 (1) | 0 (0)
Pressure ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Suspected deep tissue injury
Cellulitis of abdominal wall (Infections and infestations) | 0 (0) | 1 (1)
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Venous ulcer recurrent (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Varicose veins of lower extremities with ulcer (Vascular disorders) | 0 (0) | 1 (1)
Wound (Infections and infestations) | 0 (0) | 1 (1) — Wound in the neck of the foot

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT05892341/Prot_SAP_000.pdf